CLINICAL TRIAL: NCT04261868
Title: Virtual Reality Game Playing in Amblyopia Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamideh Sabbaghi (Other)
Responsible Party: Sponsor-Investigator, Hamideh Sabbaghi, Principal Investigator, Shahid Beheshti University of Medical Sciences
Organization: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.SBMU.ORC.REC.1398.024
Record Dates: First submitted 2020-01-30; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Dichoptic playing games with fine stimulation will present to the amblyopic eye.
  Interventions: Device: Virtual Reality
- Patching (Active Comparator): Non- amblyopic eye will be recommended to patch.
  Interventions: Other: Patching

INTERVENTIONS:
Device: Virtual Reality — New treatment for amblyopia therapy using playing games
  Other Names: No additional intervention
  Arms: Virtual Reality
Other: Patching — Patching
  Arms: Patching

SUMMARY:
Background: "Amblyopia is a neurodevelopmental disorder in both monocular and binocular functions and it extends even beyond the primary visual integration centers", therefore, amblyopia is not a "lazy eye" but it is a "lazy brain".

Purpose: The investigators aimed to compare the visual outcome of occlusion therapy with virtual reality game playing as a new therapy on amblyopic children.

Methods: This RCT was performed on 50 children with unilateral amblyopia ,4 to 10 years old. They were randomly divided to case and control (each= 25) groups. case group were trained binocularly using the virtual reality games through head set for one hour a day, 5 days in a week for 4 to 6 weeks. Controls occluded their non- amblyopic eyes, 2, 4 and 6 hours for mild (0.2 to 0.3 LogMAR), moderate (0.3 to 0.6 LogMAR) and severe (BCVA < 0.6 LogMAR) amblyopia, respectively.

ELIGIBILITY:
Inclusion Criteria:

- The best corrected visual acuity worse than 0.3 LogMAR

Exclusion Criteria:

* Patients with abnormal fixation
* Patients with neurological problems
* Patients with any types of ocular pathologies

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-03-11 (Estimated); Primary Completion 2021-05-11 (Estimated); Study Completion 2021-06-11 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | baseline and 6 months after training
  Change from baseline BCVA at 6 months

IPD SHARING:
Plan to Share IPD: Undecided